CLINICAL TRIAL: NCT03312582
Title: Efficacy of Locally Delivered 1% Metformin Gel in the Treatment of Peri-implantitis in Type2 Diabetes Mellitus Patients: A Randomized Controlled Clinical Trial
Brief Title: Locally Delivered 1% Metformin Gel in Peri-implantitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Zohaib Akram, Director, Clinical Research, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FR-17-75
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual debridement and 1% metformin gel (Experimental)
  Interventions: Drug: 1% local metformin gel
- Manual debridement and placebo (Placebo Comparator)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Drug: 1% local metformin gel — After providing manual debridement in deep peri-implant probing depths, 1% metformin gel will be applied.
  Arms: Manual debridement and 1% metformin gel
Procedure: Placebo
  Other Names: After providing manual debridement in deep peri-implant probing depths, placebo gel will be applied.
  Arms: Manual debridement and placebo

SUMMARY:
This study evaluates the efficacy of 1% local metformin gel in deep periimplant pockets of type 2 diabetes mellitus patients. Half of the participants will receive 1% metformin gel with manual debridement while the other half will receive a placebo with manual debridement.

DETAILED DESCRIPTION:
Metformin is an oral hypoglycemic drug categorized under biguanide and are considered the most efficient agents widely used in the treatment of type 2 diabetes mellitus.The general clinical benefits observed in therapy with MF seem to be greater than expected. They induce osteoblast cells to promote early bone formation through AMP kinase (AMPK) activity. Moreover, in a recent in vitro study, MF facilitated in the proliferation of MG63 osteoblast like cells. Thus, their action in stimulating bone formation has justified their use in the treatment of perimplantitis.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients.
* Patients with peri-implantitis

Exclusion Criteria:

* History of any other systemic diseases
* Cigarette smokers
* Smokeless tobacco users
* Patients who underwent scaling in the last 1 year
* Patients who took antibiotics in tje past 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2016-08-14 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | 6 months
  Marginal bone loss will be assessed on digital radiographs on calibrated computer screen.
Peri-implant prpbing depth | 6 months
  Will be measured with UNC-15 periodontal probe from crest of the gingival margin to the base of the peri-implant probing depth.

IPD SHARING:
Plan to Share IPD: Undecided